CLINICAL TRIAL: NCT01707862
Title: Surgical Management of Intravenous Leiomyomatosis With Intracardiac Extension: Our Experience and Outcomes
Brief Title: Surgery for Intravenous Leiomyomatosis
Acronym: SIVL
Status: Completed | Type: Observational
Sponsor: Li Yang (Other)
Responsible Party: Sponsor-Investigator, Li Yang, Doctor, General Hospital of Beijing PLA Military Region
Organization: General Hospital of Beijing PLA Military Region (Other)
Other Study IDs: GHBeijing-20121012
Record Dates: First submitted 2012-10-14; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Leiomyomatosis
Keywords: Intravenous leiomyomatosis; Surgery; Smooth muscle tumor
MeSH Terms: conditions — Leiomyomatosis; Smooth Muscle Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Intravenous leiomyomatosis (IVL) with intracardiac extension is a rare benign smooth muscle tumor. Reviewing literature, intracardiac extension of the IVL has been reported in at least 70 cases. Most are individual case reports. Surgical experience is not much. However, different opinion of surgical strategies remain controversial. The purpose of this report is to describe our experience of surgical management for the IVL with intracardiac extension.

DETAILED DESCRIPTION:
All patients underwent surgical management. Clinical data were obtained from medical reports. Following-up was made through email and telephone.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years.
* Tumor markers were all within normal limits.
* Patients underwent surgical management.
* Patients were followed-up for more than 12 months.

Exclusion Criteria:

-Tumor markers were all within abnormal limits

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From March 1997 to June 2011, 6 women patients were admitted to our hospital with intravenous leiomyomatosis with intracardiac extension.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 1997-03; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Genetal Hospital Beijing Military Region, First class, Principal Investigator — Institute of Cardiovascular Disease
Locations (1):
- Institute of Cardiovascular Disease, Beijing, China